CLINICAL TRIAL: NCT01992900
Title: A Phase II, Open-label, Multicentre, Pharmacokinetic, Pharmacodynamics and Safety Study of a New Paediatric Eurartesim Dispersible Formulation and Crushed Film Coated Eurartesim Tablet, in Infant Patients With P. Falciparum Malaria
Brief Title: A Pharmacokinetic/Pharmacodynamic Study of Eurartesim Dispersible Formulation in Infants With P.Falciparum Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST3073-ST3074-DM-12-002; 2013-002255-15 (EudraCT Number)
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Malaria,Falciparum
Keywords: Plasmodium falciparum Malaria; Eurartesim; ACT
MeSH Terms: conditions — Malaria, Falciparum | interventions — artenimol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eurartesim dispersible oral tablets (Experimental): Each patient will receive a specific amount of drug according to his/her body weight, once a day for three consecutive days (from 5 to <7 kg: 1 tablet containing 80 mg PQP and 10 mg DHA; from 7 to < 13 kg: 1 tablet containing 160 mg PQP and 20 mg DHA).
  Interventions: Drug: Eurartesim dispersible oral tablet
- Eurartesim film coated tablet (Active Comparator): Each patient will receive a specific amount of drug according to his/her body weight, once a day for three consecutive days (from 5 to <7 kg: half tablet equal to 80 mg PQP and 10 mg DHA; from 7 to < 13 kg: 1 tablet containing 160 mg PQP and 20 mg DHA).
  Interventions: Drug: eurartesim film coated tablet

INTERVENTIONS:
Drug: Eurartesim dispersible oral tablet — The first dose of Eurartesim dispersible oral tablet will be administered immediately after randomization. the other two doses will be administered with an interval of 24 hours. Eurartesim tablet will be dispersed in about 10 mL of water.
  Other Names: Piperaquine tetraphosphate plus dihydroartemisinin
  Arms: Eurartesim dispersible oral tablets
Drug: eurartesim film coated tablet — The first dose of Eurartesim film coated tablet will be administered immediately after randomization. the other two doses will be administered with an interval of 24 hours. tablet will be crushed and dispersed in a few amount of water (about 10 ml).
  Other Names: Piperaquine tetraphosphate plus dihydroartemisinin
  Arms: Eurartesim film coated tablet

SUMMARY:
There is a need for paediatric formulations that permit accurate dosing and enhance patient compliance. However, for the treatment of malaria, scarce paediatric-friendly formulations are available on the market. Thus, a new water dispersible formulation of eurartesim has been developed for oral administration.

Aim of this study is to provide data on pharmacokinetic profile, safety and efficacy of this new paediatric formulation and compare it with the crushed film coated tablet in infant patients (6 to ≤12 months of age) suffering from uncomplicated Plasmodium falciparum malaria.

Furthermore, a Pharmacokinetic/Pharmacodynamic(PK/PD) modelling will be built up to establish PK/PD relationship in adult and paediatric populations.

DETAILED DESCRIPTION:
Although the significant advances made during the last decades in controlling malaria in Africa, morbidity and mortality in sub-Saharan countries remain substantial. It is estimated that around 655.000 deaths a year still occur due to malaria infection and the majority of such deaths occur among young African children.

In response to the emergence and spread of classical drug-resistant Plasmodia strains, the WHO recommends since 2004 the use of artemisinin-based combination therapies (ACTs) in the treatment of uncomplicated malaria episodes.

The artemisinin derivatives are currently the most rapidly acting and potent antimalarial drugs.

Eurartesim is a fixed-dose combination product composed of dihydroartemisinin (DHA) and piperaquine phosphate (PQP). This second compound assures the long-term efficacy of eurartesim completing the whole body cleaning from the parasites. Eurartesim appears to offer benefits over existing licensed malaria treatments and is in line with current WHO treatment policy recommendations.

Eurartesim obtained a centralized marketing authorization by the European Union as film coated tablets containing 160 mg PQP/20 mg DHA and 320 mg PQP/40 mg DHA. The drug, licensed for its use in children (above 6 months of age) and adults has been administered in infants (above 6 months) and young children by crushing the tablets and administering them with a small amount of water.

According to the Guidelines on Clinical Investigation of Medicinal Products in the Paediatric Population (EMA ICH Topic E 11), there is a need for paediatric formulations that permit accurate dosing and enhance patient compliance.

However, for the treatment of malaria, scarce paediatric-friendly formulations are available on the market, and this is a particularly blatant problem as young children carry the brunt of the malaria burden. Thus, a new water dispersible formulation of eurartesim has been developed for oral administration, since liquid formulations may be needed or desirable for paediatric patients of smaller ages due to their inability to swallow tablets. Moreover, in order to increase paediatric compliance to treatment, the new formulation is prepared with acceptable flavour and sweetener for children.

Eurartesim is a promising effective ACT treatment for malaria. It provides a simple dosing scheme (a single daily dose over 3 days) and it does not need any concomitant administration of food to improve its absorption. Moreover, eurartesim offers an interesting post-treatment prophylactic effect following therapy, reducing the risk of new infection, an issue of particular relevance in highly endemic malaria countries.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female infants aged from 6 months to ≤ 12 months included.
* Ability to swallow oral suspension.
* Body weight >5 kg.
* Uncomplicated malaria, with microscopically confirmed mono-infection by P. falciparum (parasitaemia ≥1000/microL and <200000/microL).
* History of fever anytime during the preceding 48 hours or presence of fever (axillary temperature ≥37.5 °C or ≥38.0 °C rectally).
* Ability of parents or guardians to understand the nature of the trial and providing signed informed consent.
* Stable residence in the study area during the two months after recruitment and willingness to comply with the study protocol and the study visit schedule.

Exclusion Criteria:

* Antimalarial treatment with amodiaquine, chloroquine, quinine or lumefantrine-based compounds within the previous 6 weeks, with piperaquine-based compound, or mefloquine, or sulphadoxine pyrimethamine within the previous 3 months and with halofantrine within the 30 days prior to screening.
* Any other antimalarial treatment or antibiotics with antimalarial activity (including cotrimoxazol) and any herbal products, within the 7 days prior to screening.
* Severe malnutrition (defined as weight for height <70% of the median National Center for Health Statistics(NCHS)/WHO reference).
* Severe vomiting or dehydration.
* Presence of jaundice.
* Known hypersensitivity to the artemisinin-based therapy or piperaquine.
* History of relevant clinical allergic reaction of any origin.
* Clinical and/or laboratory features of severe malaria.
* Known moderate/ severe renal or liver insufficiency.
* Evidence of clinically relevant haematological, pulmonary, metabolic-endocrine, neurological, urogenital diseases as judged by the investigator.
* Already diagnosed HIV infection, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Previous admission for, or evidence of symptomatic cardiac arrhythmias or with clinically relevant bradycardia at screening (bpm < 90).
* Family history of sudden death, or known congenital prolongation of the QT interval, or any clinical condition known to prolong the QT interval.
* ECG abnormality that requires urgent management.
* Any treatment which can induce a lengthening of QT interval.
* Gastrointestinal dysfunction that could alter absorption or motility (i.e. malabsorption syndromes, intestinal sub-occlusion or previous major gastrointestinal surgery).
* Any contraindication to blood sampling.
* Moderate and severe anaemia (Hb < 7 g/dL).
* Patients who have used any drugs or substances known to be strong inhibitors of Cytochrome P enzymes (formerly known as cytochrome P450 enzymes) within 10 days prior to screening.
* Patients who have used any drugs or substances known to be strong inducers of CYP enzymes (formerly known as cytochrome P450 enzymes)within 28 days prior to screening.
* Children lactated by HIV positive women who are undergoing treatment with antiretroviral drugs.
* Participation in any investigational drug study during the 30 days prior to screening or previously randomised in the present trial.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Comparison of peak plasma concentration of Dihydroartemisinin in the two studied formulations | DHA plasma samples will be collected on the first day of study drug administration at 20, 30, 40, 60, 100, 200 and 300 minutes post-dose
  In order to minimize the blood sampling in infants, patients will be divided into 10 blood sampling groups for both the treatments (water dispersible and crushed film coated tablet) and only 2 blood draws per group will be taken within the prespecified timepoints.
  Optimal sampling design was performed by using the appropriate software. The D-optimal design option was used to determine the optimal sampling design.
Comparison of area under the plasma concentration versus time curve of Dihydroartemisinin in the two studied formulations. | DHA plasma samples will be collected on the first day of study drug administration at 20, 30, 40, 60, 100, 200 and 300 minutes post-dose
  In order to minimize the blood sampling in infants, patients will be divided into 10 blood sampling groups for both the treatments (water dispersible and crushed film coated tablet) and only 2 blood draws per group will be taken within the pre-specified timepoints.
  Optimal sampling design was performed by using the appropriate software. The D-optimal design option was used to determine the optimal sampling design.
Comparison of peak plasma concentration of Piperaquine in the two studied formulations | PQP plasma samples will be collected on day 0 of treatment at 40, 80, 280, 720 minutes, then on day 1 at 24 hours and on day 2 at 40, 80, 280, 720 minutes after the last drug administration and then 24, 120, 288 and 456 hours
  In order to minimize the blood sampling in infants, patients will be divided into 10 blood sampling groups for both the treatments (water dispersible and crushed film coated tablet) and only 2 blood draws per group will be taken within the pre-specified timepoints.
  Optimal sampling design was performed by using the appropriate software. The D-optimal design option was used to determine the optimal sampling design.
Comparison of area under the plasma concentration versus time curve of Piperaquine in the two studied formulations. | PQP plasma samples will be collected on day 0 of treatment at 40, 80, 280, 720 minutes, then on day 1 at 24 hours and on day 2 at 40, 80, 280, 720 minutes after the last drug administration and then 24, 120, 288 and 456 hours
  In order to minimize the blood sampling in infants, patients will be divided into 10 blood sampling groups for both the treatments (water dispersible and crushed film coated tablet) and only 2 blood draws per group will be taken within the pre-specified timepoints.
  Optimal sampling design was performed by using the appropriate software. The D-optimal design option was used to determine the optimal sampling design.

SECONDARY OUTCOMES:
Parasite clearance time | At screening and then about every 12 hours until the time of the first negative result, then confirmed by a second negative result or up to three days
  Blood film for parasite count will be read by two independent microscopists.
Fever clearance time | At screening and then about every 12 hours until the time on which body temperature falls down below 37.5 °C, or up to three days
  Body temperature will be recorded to collect information about the fever clearance time
Change from baseline of electrocardiographic QT interval at 4-6 hours after the last study drug intake | Before randomization and then at 4-6 hours after the last dose of study drug.
  Triplicate ECGs will be undertaken on screening (before study drug administration)as well as 4-6 hours after the last drug administration.
  The triplicate ECG values will be averaged in order to obtain one single value per patient and time point. These averages will be used for the statistical analysis.
  From the collected values the heart rate corrected QT intervals will be derived according to Fridericia's correction (QTcF)
Blood chemistry: proportion of patients with deterioration of parameters at day 7 respect to screening. | screening and Day 7
  The evaluated analytes are: Blood Urea Nitrogen, Creatinine, Glucose, Alanine aminotransferase, aspartate aminotransferase, Total Bilirubin, electrolytes (Na+, K+ and Cl-)
Hematology: proportion of patients with deterioration of parameters at day 7 respect to screening | screening and day 7
  the following parameters are evaluated: Hemoglobin, hematocrit and full blood counts including Red Blood Cell and differential White Blood Cells, Platelet Count
Adverse Events occurrence to calculate percentage of patients experiencing Adverse Events and Serious Adverse Events | during all the study period from randomization and up to day 42

CONTACTS AND LOCATIONS:
Overall Officials: Enrique O Bassat, MD, Study Chair — Manica's health Research Centre, centre de investigacao Saude-Manica (CISM)
Locations (7):
- Burkina Faso (2):
  - Centre Muraz, Bobo-Dioulasso
  - Centre National de Recherche et de Formation en Paludisme, Ouagadougou
- Kinshasa School of Public Health, School of Medicine, University of Kinshasa, Kinshasa, Democratic Republic of the Congo
- Manica's Health Research Centre, Manica, Mozambique
- Tanzania (2):
  - Bagamoyo Research center, Ifakara Heath Institute, Bagamoyo
  - National Insititute for Medical Research, Tanga
- Medical Research Council, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Belard S, Ramharter M, Kurth F. Paediatric formulations of artemisinin-based combination therapies for treating uncomplicated malaria in children. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD009568. doi: 10.1002/14651858.CD009568.pub2. PMID 33289099
- [Derived] Gargano N, Madrid L, Valentini G, D'Alessandro U, Halidou T, Sirima S, Tshefu A, Mtoro A, Gesase S; Eurartesim Dispersible Study Group; Bassat Q. Efficacy and Tolerability Outcomes of a Phase II, Randomized, Open-Label, Multicenter Study of a New Water-Dispersible Pediatric Formulation of Dihydroartemisinin-Piperaquine for the Treatment of Uncomplicated Plasmodium falciparum Malaria in African Infants. Antimicrob Agents Chemother. 2017 Dec 21;62(1):e00596-17. doi: 10.1128/AAC.00596-17. Print 2018 Jan. PMID 29061746